CLINICAL TRIAL: NCT03617653
Title: EaRneST: Exercise and CiRulating MetabolomicS: A Pilot Randomized Controlled Study
Acronym: EaRneST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018/2118
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Disease Other
MeSH Terms: interventions — Chromosomes, Human, 1-3; Walk Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Intervention (Other): Baseline procedure, Bio specimen collection , Six minute walk, Musculoskeletal Analysis, Exercise intervention from Visit 2 to Visit 13, End of 3 month assessment.
  Interventions: Diagnostic Test: Group A
- Group B- Control (Other): Baseline procedure, Bio specimen collection , Six minute walk, Musculoskeletal Analysis & End of 3 month assessment.
  Interventions: Diagnostic Test: Group A

INTERVENTIONS:
Diagnostic Test: Group A — Refer to detailed study Description
  Other Names: six minute walk test; exercise intervention

SUMMARY:
Brief Summary The purpose of this study is to investigate how circulating metabolites mediate changes in heart function after exercise intervention.

Condition or disease :Cardiovascular function

Intervention/treatment Cardiovascular: Echocardiography Other: Vascular Stiffness Other: Metabolomics (Blood)

DETAILED DESCRIPTION:
Detailed Description The purpose of the study is to determine the effect of a structured exercise intervention on mitochondrial fuel metabolism and cardiovascular function. Participants with diastolic dysfunction will undergo a structured exercise intervention.

Group A (intervention) will undergo exercise intervention for three months and Group B (control) will not receive the exercise intervention. At the start of the study and upon completion, all participants will undergo cardiovascular tests to measure cardiovascular function, as well bio-specimen (blood and urine) collection for metabolic profiling.

Study Design Study Type : Randomized controlled trial Estimated Enrollment :40 participants Time Perspective:Prospective Official Title:EaRneST: Exercise and CiRculating MetabolomicS: A Pilot Randomized Controlled Study Study Start Date :July 2018 Estimated Primary Completion Date :Nov 2019 Estimated Study Completion Date : Nov 2019

Groups and Cohorts Group/Cohort :Group A Intervention/treatment Visit 1. Baseline procedures

1. Cardiovascular measurements Arterial stiffness assessment by non-invasive brachial blood pressure machine Echocardiography Standard transthoracic echocardiographic examination will be performed according to established laboratory practice using standard commercially available machines.

   Resting electrocardiography will be performed to ascertain sinus rhythm.
2. Biospecimen collection Fresh blood, urine specimens will be collected for metabolomics.
3. Six-minute walk test The Six-Minute Walk Test is a shuttle walk test.
4. Musculoskeletal Analysis Participants will undergo focused examinations that include measurement of height, weight, body mass index, waist circumference, body composition analysis.

Visit 2 to Visit 13. One time per week exercise intervention for a total of three months

Visit 14: End of three months' procedures.

1. Cardiovascular measurements Echocardiography Resting electrocardiography will be performed to ascertain sinus rhythm.
2. Biospecimen collection Fresh blood, urine specimens will be collected for metabolomics.
3. Six-minute walk test
4. Musculoskeletal Analysis

Group B Visit 1. Baseline procedures

1. Cardiovascular measurements Arterial stiffness assessment by non-invasive brachial blood pressure machine Echocardiography Standard transthoracic echocardiographic examination will be performed according to established laboratory practice using standard commercially available machines.

   Resting electrocardiography will be performed to ascertain sinus rhythm.
2. Biospecimen collection Fresh blood, urine specimens will be collected for metabolomics.
3. Six-minute walk test The Six-Minute Walk Test is a shuttle walk test.
4. Musculoskeletal Analysis Participants will undergo focused examinations that include measurement of height, weight, body mass index, waist circumference, body composition analysis.

Visit 2: End of three months' procedures.

1. Cardiovascular measurements Arterial stiffness assessment by non-invasive brachial blood pressure machine Echocardiography Resting electrocardiogram will be performed to ascertain heart rhythm.
2. Biospecimen collection Fresh blood, urine specimens will be collected for metabolomics.
3. Six-minute walk test
4. Musculoskeletal Analysis Outcome Measures

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years old and above
* At least Grade 1 Diastolic Dysfunction
* Willing and able to give informed consent for participation for the study

Exclusion Criteria:

* History of cardiovascular disease
* History of cancer
* History of stroke
* Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥90mmHg) despite being on treatment for hypertension
* Low blood pressure (systolic blood pressure <90mmHg or diastolic blood pressure <40mmHg)
* Acute pulmonary embolus or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or known dissecting aneurysm
* Acute systemic infection
* Uncontrolled metabolic disease (e.g. diabetes, thyrotoxicosis or myxedema)
* Neuromuscular, musculoskeletal or rheumatoid disorders that are exacerbated by exercise

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Metabolmic Profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Su-Mei Angela Koh, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wong JJ, Ho JS, Teo LLY, Wee HN, Chua KV, Ching J, Gao F, Tan SY, Tan RS, Kovalik JP, Koh AS. Effects of short-term moderate intensity exercise on the serum metabolome in older adults: a pilot randomized controlled trial. Commun Med (Lond). 2024 May 4;4(1):80. doi: 10.1038/s43856-024-00507-w. PMID 38704414